CLINICAL TRIAL: NCT01019356
Title: Role of Insulin Action and Free Fatty Acids in Hyperandrogenism and Role of Metabolism of Inositols in Insulin Resistance of Women With Polycystic Ovary Syndrome
Brief Title: Role of Insulin Action and Free Fatty Acids in Hyperandrogenism of Women With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jean-Patrice Baillargeon (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor-Investigator, Jean-Patrice Baillargeon, MD, Université de Sherbrooke
Organization: Université de Sherbrooke (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 06-075
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Polycystic Ovary Syndrome
Keywords: PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Rosiglitazone; Acarbose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rosiglitazone (Experimental): Lean and obese PCOS women
  Interventions: Drug: Rosiglitazone
- Acarbose (Active Comparator): Obese PCOS women
  Interventions: Drug: Acarbose
- Control (No Intervention): Obese and lean healthy women evaluated only at baseline

INTERVENTIONS:
Drug: Rosiglitazone — 4 mg twice daily for 8 weeks orally
  Other Names: Avandia
  Arms: Rosiglitazone
Drug: Acarbose — 100 mg three times daily for 8 weeks orally
  Other Names: Prandase
  Arms: Acarbose

SUMMARY:
The investigators hypothesis is that free fatty acids (FFA) accumulation in non fatty tissues would lead to insulin resistance and hyperandrogenism in PCOS women. Accordingly, Peroxisome Proliferator-Activated Receptor gamma (PPARγ) agonist (rosiglitazone) would be a great therapeutic option for PCOS as their activation induces transcription factors of gene implicated in fatty acids metabolism.

The aim is to verify if insulin-related hyperandrogenism can be reversed in women having polycystic ovary syndrome following an 8-week treatment with rosiglitazone compared to simple insulin reduction with acarbose.

For the purpose of this study, 14 lean women (BMI ≤ 25 kg/m2) and 36 obese women (BMI 30-39 kg/m2) with PCOS as well as 14 lean and 14 obese control women will be recruited to determine their insulin sensibility (insulin levels, M-value, metabolic clearance rate of glucose)and FFA metabolism (FFA levels, rythm of apparition and disapearance of FFA) during a 75g oral glucose tolerance test and a 2-step insulin-glucose clamp.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very common but complex endocrine disorder affecting 6 to 10% of childbearing age women. To diagnose PCOS, women must display two of these three symptoms: clinical or biochemical hyperandrogenism, oligoamenorrhea, and/or echographycally confirmed polycystic ovary. Many studies have also demonstrated that PCOS women are more insulin resistant than control women when matched for body mass index (BMI). Thus, insulin resistance (IR) and secondary hyperinsulinemia would be important premises in the development of PCOS. In fact, the prevalence of type 2 diabetes (T2D) is tripled in PCOS women.

Higher free fatty acid (FFA) concentrations were also observed in the circulation of PCOS women. As FFA accumulates in liver and muscle instead of fat cells, this could be an important cause of IR according to the theory of lipotoxicity. Some indirect evidences are suggesting that FFA accumulation in androgen secreting cells (ovary and adrenal gland) could enhance their androgen production. Based on these findings, our hypothesis is that FFA accumulation in non fatty tissues would lead to IR and hyperandrogenism in PCOS women. Accordingly, Peroxisome Proliferator-Activated Receptor gamma (PPARγ) agonist (rosiglitazone) would be a great therapeutic option for PCOS as their activation induces transcription factors of gene implicated in fatty acids metabolism.

The aim is to verify if insulin-related hyperandrogenism can be reversed in PCOS women following an 8-week treatment with rosiglitazone compared to simple insulin reduction with acarbose. For the purpose of this study, 14 lean women (BMI ≤ 25 kg/m2) and 36 obese women (BMI 30-39 kg/m2) with PCOS as well as 14 lean and 14 obese control women will be recruited to determine their insulin sensibility (insulin levels, M-value, metabolic clearance rate of glucose)and FFA metabolism (FFA levels, rythm of apparition and disapearance of FFA) during a 75g oral glucose tolerance test and a 2-step insulin-glucose clamp.

ELIGIBILITY:
Inclusion Criteria:

PCOS :

* Biochemical hyperandrogenism (free testosterone ≥ 50 pmol/l)
* Oligomenorhea (≤ 8 menstrual cycle per year)

Health volunteers :

* Normal menstrual cycle
* Normal levels of free and total testosterone
* No family history with PCOS

Exclusion Criteria:

* Diabetes or glucose intolerance
* Current or past use within 3 months of oral contraceptives
* Current or past use within 3 months of medications known to affect insulin sensitivity (metformin, PPARy agonists, b-blockers, thiazides, calcium channel blockers, glucocorticoids, etc.)
* Pulmonary, cardiac, renal, hepatic, neurologic, psychiatric, infectious or neoplastic disease (other than non-melanoma skin cancer)
* Documented or suspected recent (within one year) history of drug abuse or alcoholism
* Use of any investigational drug within three months prior to study onset

Healthy volunteers :

* History of gestational diabetes
* Positive family history for first-degree relative with diabetes
* Disorders linked to insulin resistance (hypertension, dyslipidemia or acanthosis nigricans)

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2006-08; Primary Completion 2021-07 (Actual); Study Completion 2021-07 (Actual)

PRIMARY OUTCOMES:
Androgen hyper-responsiveness to insulin - Ratio | 8 weeks
  The calculated ratio of free testosterone to the area under the insulin curve during an OGTT

SECONDARY OUTCOMES:
Androgen hyper-responsiveness to insulin - Relationship | 8 weeks
  Determined by the relationship between testosterone and insulin levels during an OGTT.
Insulin sensitivity | 8 weeks
  Determined by a 2-step insulin-glucose clamp
Insulin secretion | 8 weeks
  Determined by a 2-step insulin-glucose clamp
Hepatic glucose production | 8 weeks
  Determined by a 2-step insulin-glucose clamp
Plasma DCI-IPG during euglycemic-hyperinsulinemic clamp | 8 weeks
  Measured during steady-state

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Patrice Baillargeon, MD, MSc, Principal Investigator — Université de Sherbrooke
Locations (1):
- Université de Sherbrooke, Sherbrooke, Quebec, Canada